CLINICAL TRIAL: NCT01330459
Title: An Evaluation of Hydrocodone/Acetaminophen for Pain Control in First Trimester Surgical Abortion
Brief Title: Hydrocodone For Pain Control in First Trimester Surgical Abortion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Elizabeth Micks (Other)
Collaborators: Planned Parenthood Federation of America (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Micks, Fellow in Family Planning, Oregon Health and Science University
Organization: Oregon Health and Science University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OHSU FAMPLAN 6734
Record Dates: First submitted 2011-04-01; First posted 2011-04-07 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Pain
Keywords: Pain during first trimester surgical abortion
MeSH Terms: conditions — Pain | interventions — oxycodone-acetaminophen; acetaminophen, hydrocodone drug combination; Ibuprofen; Lorazepam; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrocodone/acetaminophen (Active Comparator): Subject will receive hydrocodone/acetaminophen 45-90 minutes prior to abortion procedure.
  Subject will also recieve ibuprofen, lorazepam, and lidocaine 45-90 minutes prior to abortion procedure.
  Interventions: Drug: Hydrocodone/acetaminophen; Drug: Ibuprofen; Drug: Lorazepam; Drug: Lidocaine
- Placebo (Placebo Comparator): Subject will receive placebo 45-90 minutes prior to abortion procedure.
  Subject will also recieve ibuprofen, lorazepam, and lidocaine 45-90 minutes prior to abortion procedure.
  Interventions: Drug: Placebo; Drug: Ibuprofen; Drug: Lorazepam; Drug: Lidocaine

INTERVENTIONS:
Drug: Hydrocodone/acetaminophen — Administration of 2 tablets 5/325mg hydrocodone/acetaminophen 45-90 minutes prior to procedure.
  Other Names: Vicodin
  Arms: Hydrocodone/acetaminophen
Drug: Placebo — Administration of 2 tablets methylcellulose (placebo) 45-90 minutes prior to procedure.
  Arms: Placebo
Drug: Ibuprofen — 800 mg oral ibuprofen
Drug: Lorazepam — 2 mg oral lorazepam
Drug: Lidocaine — 20 ml 1% buffered lidocaine, injected

SUMMARY:
The purpose of this study is to determine whether preoperatively administered hydrocodone/acetaminophen (HC/APAP) reduces pain during a first trimester surgical abortion.

DETAILED DESCRIPTION:
The investigators plan to conduct a double-blinded randomized placebo-controlled trial of 120 women undergoing elective first trimester surgical abortion. These women will be premedicated with either two tabs of 5/350 hydrocodone/acetaminophen or 2 tabs of a placebo. All subjects will receive ibuprofen and lorazepam preoperatively and a PCB. This study will examine the incremental benefit of HC/APAP over this standard medication regimen. Randomization will be stratified into two groups. Subjects less than 8 weeks gestation will comprise the early gestational age group. Subjects between 8 weeks 0 days and 10 weeks 6 days will comprise the late gestational age group. The investigators will be assessing patient perception of pain, nausea, satisfaction, and anxiety at multiple points during the clinic visit using 100-mm visual analogue scales (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Voluntarily requesting surgical pregnancy termination
* Pregnancy with intrauterine gestational sac up to 10 weeks 6 days gestation, dated by ultrasound
* Eligible for suction curettage
* English or Spanish speaking
* Good general health
* Able and willing to give informed consent and agree to terms of the study

Exclusion Criteria:

* Gestational ages 11 weeks or more
* Incomplete abortion
* Premedication with misoprostol
* Use of any opioid medication within the past 7 days
* Use of heroin within the past 7 days
* Requested opioids or IV sedation prior to start of the procedure
* Patients who refuse ibuprofen or lorazepam
* Contraindications or allergies to HC/APAP, lidocaine, ibuprofen, or lorazepam
* Significant medical problem necessitating inpatient procedure
* Adnexal mass or tenderness on pelvic exam consistent with pelvic inflammatory disease
* Known hepatic disease

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Micks, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Planned Parenthood CW, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Background] Allen RH, Kumar D, Fitzmaurice G, Lifford KL, Goldberg AB. Pain management of first-trimester surgical abortion: effects of selection of local anesthesia with and without lorazepam or intravenous sedation. Contraception. 2006 Nov;74(5):407-13. doi: 10.1016/j.contraception.2006.06.002. Epub 2006 Aug 2. PMID 17046383
- [Background] Belanger E, Melzack R, Lauzon P. Pain of first-trimester abortion: a study of psychosocial and medical predictors. Pain. 1989 Mar;36(3):339-350. doi: 10.1016/0304-3959(89)90094-8. PMID 2710563
- [Background] Bone ME, Dowson S, Smith G. A comparison of nalbuphine with fentanyl for postoperative pain relief following termination of pregnancy under day care anaesthesia. Anaesthesia. 1988 Mar;43(3):194-7. doi: 10.1111/j.1365-2044.1988.tb05538.x. PMID 3364636
- [Background] Dahl V, Fjellanger F, Raeder JC. No effect of preoperative paracetamol and codeine suppositories for pain after termination of pregnancies in general anaesthesia. Eur J Pain. 2000;4(2):211-5. doi: 10.1053/eujp.2000.0174. PMID 10957701
- [Background] Edelman A, Nichols MD, Jensen J. Comparison of pain and time of procedures with two first-trimester abortion techniques performed by residents and faculty. Am J Obstet Gynecol. 2001 Jun;184(7):1564-7. doi: 10.1067/mob.2001.114858. PMID 11408881
- [Background] Edelman A, Nichols MD, Leclair C, Astley S, Shy K, Jensen JT. Intrauterine lidocaine infusion for pain management in first-trimester abortions. Obstet Gynecol. 2004 Jun;103(6):1267-72. doi: 10.1097/01.AOG.0000127981.53911.0e. PMID 15172863
- [Background] Edelman A, Nichols MD, Leclair C, Jensen JT. Four percent intrauterine lidocaine infusion for pain management in first-trimester abortions. Obstet Gynecol. 2006 Feb;107(2 Pt 1):269-75. doi: 10.1097/01.AOG.0000194204.71925.4a. PMID 16449111
- [Background] Heath PJ, Ogg TW. Prophylactic analgesia for daycase termination of pregnancy. A double-blind study with controlled release dihydrocodeine. Anaesthesia. 1989 Dec;44(12):991-4. doi: 10.1111/j.1365-2044.1989.tb09206.x. PMID 2619027
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Kan AS, Ng EH, Ho PC. The role and comparison of two techniques of paracervical block for pain relief during suction evacuation for first-trimester pregnancy termination. Contraception. 2004 Aug;70(2):159-63. doi: 10.1016/j.contraception.2004.03.013. PMID 15288222
- [Background] Nichols, M. D., Halvorson-Boyd, G., Goldstein, R., Gevirtz, C., & Healow, D. (2009). Pain management. In M. Paul, E. S. Lichtenberg, L. Borgatta, D. A. Grimes & P. G. Stubblefield (Eds.), Management of unintended and abnormal pregnancy. (pp. 90-110): Wiley-Blackwell.
- [Background] O'Connell K, Jones HE, Simon M, Saporta V, Paul M, Lichtenberg ES; National Abortion Federation Members. First-trimester surgical abortion practices: a survey of National Abortion Federation members. Contraception. 2009 May;79(5):385-92. doi: 10.1016/j.contraception.2008.11.005. Epub 2008 Dec 11. PMID 19341852
- [Background] Renner RM, Jensen JT, Nichols MD, Edelman A. Pain control in first trimester surgical abortion. Cochrane Database Syst Rev. 2009 Apr 15;2009(2):CD006712. doi: 10.1002/14651858.CD006712.pub2. PMID 19370649
- [Background] Romero I, Turok D, Gilliam M. A randomized trial of tramadol versus ibuprofen as an adjunct to pain control during vacuum aspiration abortion. Contraception. 2008 Jan;77(1):56-9. doi: 10.1016/j.contraception.2007.09.008. Epub 2007 Nov 26. PMID 18082668
- [Background] Rowbotham MC. What is a "clinically meaningful" reduction in pain? Pain. 2001 Nov;94(2):131-132. doi: 10.1016/S0304-3959(01)00371-2. No abstract available. PMID 11690725
- [Background] Singh RH, Ghanem KG, Burke AE, Nichols MD, Rogers K, Blumenthal PD. Predictors and perception of pain in women undergoing first trimester surgical abortion. Contraception. 2008 Aug;78(2):155-61. doi: 10.1016/j.contraception.2008.03.011. Epub 2008 May 27. PMID 18672118
- [Background] Suprapto K, Reed S. Naproxen sodium for pain relief in first-trimester abortion. Am J Obstet Gynecol. 1984 Dec 15;150(8):1000-1. doi: 10.1016/0002-9378(84)90399-5. PMID 6507524
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Uppington, J. (2006). Opioids. In J. Ballantyne (Ed.), Massachusetts General Hospital Handbook of Pain Management (pp. 106-126). Philadelphia: Lippincott Williams & Wilkins.
- [Background] Safe Abortion: Technical and Policy Guidance for Health Systems. 2nd edition. Geneva: World Health Organization; 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK138196/ PMID 23700650
- [Background] Wiebe E, Podhradsky L, Dijak V. The effect of lorazepam on pain and anxiety in abortion. Contraception. 2003 Mar;67(3):219-21. doi: 10.1016/s0010-7824(02)00516-4. PMID 12618257
- [Background] Wiebe ER, Rawling M. Pain control in abortion. Int J Gynaecol Obstet. 1995 Jul;50(1):41-6. doi: 10.1016/0020-7292(95)02416-a. PMID 7556858
- [Derived] Micks EA, Edelman AB, Renner RM, Fu R, Lambert WE, Bednarek PH, Nichols MD, Beckley EH, Jensen JT. Hydrocodone-acetaminophen for pain control in first-trimester surgical abortion: a randomized controlled trial. Obstet Gynecol. 2012 Nov;120(5):1060-9. doi: 10.1097/aog.0b013e31826c32f0. PMID 23090523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects in this study are women 18 years or older, recruited from OHSU and PPCW who present for an elective termination of pregnancy up to 10 weeks 6 days gestation
Groups:
- Hydrocodone/Acetaminophen: Subject will receive hydrocodone/acetaminophen 45-90 minutes prior to abortion procedure.
- Placebo: Subject will receive placebo 45-90 minutes prior to abortion procedure.
Period: Overall Study
Arm/Group | Hydrocodone/Acetaminophen | Placebo
Started | 61 | 60
Completed | 61 | 58
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrocodone/Acetaminophen | Placebo | Total
Number analyzed (Participants) | 61 | 60 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 60 | 58 | 118
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.1 (6.3) | 24.7 (4.5) | 25.4 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 60 | 121
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 61 | 60 | 121

OUTCOME MEASURES:

1. Primary Outcome: Patient Perception of Pain
Description: To determine whether HC/APAP, given in addition to a standard regimen of ibuprofen, lorazepam, and PCB, affects patient pain perception at the time of uterine aspiration, as measured by distance (mm) from the left of the 100 mm visual analog scale (VAS). The number 0 indicates no pain, and 100 indicates worst pain imaginable.
Time Frame: At time of uterine aspiration (baseline)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Hydrocodone/Acetaminophen | Placebo
Number analyzed (Participants) | 61 | 58
mm | 65.7 (25.4) | 63.1 (26.6)

2. Secondary Outcome: Patient Perception of Pain During Cervical Dilation
Description: Distance (mm) from the left of the 100 mm VAS scale (VAS anchors: 0 = none, 100 mm = worst imaginable) recorded after cervical dilation
Time Frame: During procedure (approximately 45-90 min after hydrocodone/acetaminophen or placebo, and within 5 minutes of procedure starting)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Hydrocodone/Acetaminophen | Placebo
Number analyzed (Participants) | 59 | 58
mm | 47.2 (26.8) | 43.9 (28.9)

3. Secondary Outcome: Satisfaction With Pain Control
Description: Distance (mm) from the left of the 100 mm VAS (VAS anchors: 0 = unsatisfied, 100 mm = very satisfied) recorded 30 minutes after completion of the procedure.
Time Frame: 30 minutes after completion of the procedure (which started 45-90 minutes after study drug administration)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Hydrocodone/Acetaminophen | Placebo
Number analyzed (Participants) | 61 | 60
mm | 74.8 (24.7) | 67.3 (24.7)

4. Secondary Outcome: Postoperative Nausea
Description: To assess whether HC/APAP is associated with nausea, measured on the 100 mm VAS, recorded 30 minutes postoperatively. VAS anchors: 0 indicates no pain, and 100 indicates worst pain imaginable.
Time Frame: 30 minutes after completion of the procedure (which started 45-90 minutes after study drug administration)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Hydrocodone/Acetaminophen | Placebo
Number analyzed (Participants) | 60 | 58
mm | 19.4 (27.0) | 11.4 (21.5)

5. Secondary Outcome: Need for Additional Intraoperative and/or Postoperative Pain Medication
Description: To assess need for additional intraoperative and/or postoperative pain medication
Time Frame: 30 minutes after completion of the procedure (which started 45-90 minutes after study drug administration)
Measure: Count of Participants; unit: Participants
Groups:
- Hydrocodone/Acetaminophen: Subject will receive hydrocodone/acetaminophen 45-90 minutes prior to abortion procedure.
  Subject will also recieve ibuprofen, lorazepam, and lidocaine 45-90 minutes prior to abortion procedure.
  Hydrocodone/acetaminophen: Administration of 2 tablets 5/325mg hydrocodone/acetaminophen 45-90 minutes prior to procedure.
  Ibuprofen: 800 mg oral ibuprofen
  Lorazepam: 2 mg oral lorazepam
  Lidocaine: 20 ml 1% buffered lidocaine, injected
- Placebo: Subject will receive placebo 45-90 minutes prior to abortion procedure.
  Subject will also recieve ibuprofen, lorazepam, and lidocaine 45-90 minutes prior to abortion procedure.
  Placebo: Administration of 2 tablets methylcellulose (placebo) 45-90 minutes prior to procedure.
  Ibuprofen: 800 mg oral ibuprofen
  Lorazepam: 2 mg oral lorazepam
  Lidocaine: 20 ml 1% buffered lidocaine, injected
Arm/Group | Hydrocodone/Acetaminophen | Placebo
Number analyzed (Participants) | 61 | 60
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Hydrocodone/Acetaminophen | Placebo
Serious Adverse Events (participants affected / at risk) | 1/61 | 1/60
Other Adverse Events (participants affected / at risk) | 2/61 | 1/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocodone/Acetaminophen (N=61) | Placebo (N=60)
Uterine perforation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Hematometra requiring reaspiration (Reproductive system and breast disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocodone/Acetaminophen (N=61) | Placebo (N=60)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No